CLINICAL TRIAL: NCT00032929
Title: Double-Blind, Placebo-Controlled Trial of Selegiline Transdermal System for the Treatment of Cocaine Dependence
Brief Title: Selegiline Transdermal System for the Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Somerset Pharmaceuticals (Industry)
Responsible Party: Liza Gorgon, National Institute on Drug Abuse
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-CSP-1019-1; NCT00007553 (obsolete NCT alias); NCT00024700 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-05

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Selegiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Selegiline

SUMMARY:
The purpose of this study is to evaluate the Selegiline Transdermal System for the treatment of cocaine dependence.

DETAILED DESCRIPTION:
The study objectives are to assess the efficacy and safety of the Selegiline Transdermal System (STS) in reducing cocaine use in subjects with cocaine dependence. It is hypothesized that selegiline treatment compared to placebo, will be associated with fewer days of cocaine use as assessed by self-report confirmed with urine assays for benzoylecgonine (BE).

ELIGIBILITY:
Inclusion Criteria:

* Male/Female
* At least 18 years of age
* DSM-4 diagnosis of cocaine dependence
* Ability to understand and provide written consent
* Female subjects must use acceptable birth control

Exclusion Criteria:

- Additional Criteria available during the screening process at the site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2001-03; Primary Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Weekly mean proportion of cocaine non-use days
Measured reductions in cocaine and other drug use

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkashef, MD, Study Chair — National Institute on Drug Abuse (NIDA)
Locations (16):
- United States (16):
  - Tucson VA Medical Center, Tucson, Arizona
  - Haight-Ashbury Free Clinic, Berkeley, California
  - Friends Research Institute-2, Los Angeles, California
  - Friends Research Institute, Los Angeles, California
  - San Francisco General Hosptial, San Francisco, California
  - San Francisco VA Medical Center, San Francisco, California
  - Denver VA Medical Center, Denver, Colorado
  - New Orleans VA Medical Center, New Orleans, Louisiana
  - VA Maryland Healthcare System, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - VA North Texas Health Care System, Dallas, Texas
  - University of Texas Hlth Sci Ctr Houston, Houston, Texas
  - Salt Lake City VA Medical Center, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington

REFERENCES:
- [Result] Elkashef A, Fudala PJ, Gorgon L, Li SH, Kahn R, Chiang N, Vocci F, Collins J, Jones K, Boardman K, Sather M. Double-blind, placebo-controlled trial of selegiline transdermal system (STS) for the treatment of cocaine dependence. Drug Alcohol Depend. 2006 Dec 1;85(3):191-7. doi: 10.1016/j.drugalcdep.2006.04.010. Epub 2006 May 30. PMID 16730924